CLINICAL TRIAL: NCT01737047
Title: A Prospective, Observational Study to Examine the Effects of Ageing on the Clinical Outcomes of People Living With HIV in England and Ireland
Brief Title: The Effects of Ageing on the 'Pharmacokinetic and Clinical Observations in People Over Fifty'
Acronym: POPPY
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Gilead Sciences (Industry); Janssen, LP (Industry); ViiV Healthcare (Industry); Bristol-Myers Squibb (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CRO: 1992; 2012-003581-40 (EudraCT Number)
Record Dates: First submitted 2012-11-01; First posted 2012-11-29 (Estimated); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: HIV Positive; Ageing
Keywords: HIV; Ageing
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for storage Blood (serum and plasma,) and urine samples will be collected at visits 1 and 3 stored for subsequent projects of the potential pathogenic mechanisms underlying age-related diseases. This will include assessment of vitamin-D and PTH and probably DNA analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV positive over 50 years of age: All study subjects will undergo a whole body DEXA scan (dual energy X-ray absorptiometry). at the beginning and end of the study.
  Blood sample collections for the determination of the plasma concentrations of tenofovir and the third agent (i.e. a non-nucleoside reverse transcriptase, protease, entry or integrase inhibitor) in the patient's regimen will be drawn
- HIV positive under the age of 50: All study subjects will undergo a whole body DEXA scan (dual energy X-ray absorptiometry). at the beginning and end of the study.
  Blood sample collections for the determination of the plasma concentrations of tenofovir and the third agent (i.e. a non-nucleoside reverse transcriptase, protease, entry or integrase inhibitor) in the patient's regimen will be drawn
- HIV negative over the age of 50: All study subjects will undergo a whole body DEXA scan (dual energy X-ray absorptiometry). at the beginning and end of the study.

SUMMARY:
The purpose of this study is to identify medical conditions that may cause particular problems to individuals receiving care for HIV infection over the age of 50. In addition, as the effects and potentially the side effects, of HIV medication may change with age, this study will also investigate the association between age and differing effects of antiretroviral therapies such as treatment outcomes, side effects and the levels of drugs in blood.

Results from this study may inform future HIV treatment guidelines on how individuals with HIV infection are monitored. The results may also assist in the design of future studies for the treatment of diseases associated with ageing.

DETAILED DESCRIPTION:
Multicentre, prospective, observational study over 3 years.

The study will describe the impact of advancing age on the experience of living with HIV in England and Ireland. To address this cohorts of HIV-positive people aged >50 and <50 years (as well as demographically matched HIV-negative people aged >50 years) will be established.

1. To analyse the incidence and outcomes of co-morbidities in older-HIV-positive people and their relationship with demographic/clinical factors.
2. To evaluate associations between antiretroviral drug concentrations and age, and to assess the potential impact of age on drug efficacy, drug-drug interactions and co-morbidities.
3. To contribute to the development and implementation of evidence-based recommendations for the clinical monitoring of older HIV-positive patients.

2000 will be recruited in all either white or black african individuals (self reported) 1000 will be Over 50 years of age and HIV positive, 500 will be under the age of 50 and will be HIV positive and 500 will be over the age of 50 and be HIV negative.

ELIGIBILITY:
Inclusion Criteria:

Older HIV-positive cohort (n=1000):

* documented HIV infection
* age >50 years at study entry
* self defined white or black African ethnicity
* likely route of HIV acquisition via sexual exposure Either by male to male exposure if white or by heterosexual exposure if white or black African
* able to comprehend study patient information leaflet

  -Younger HIV-positive cohort (n=500):
* documented HIV infection
* age <50 at study entry*
* self defined white or black African ethnicity
* likely route of HIV acquisition via sexual exposure Either by male to male exposure if white or by heterosexual exposure if white or black African.
* able to comprehend study patient information leaflet

  * this group will comprise of at least 150 subjects in each of the following age groups: 20-29, 30-39, 40-49 years. Recruitment will be monitored by the Study Monitoring Team.

HIV-negative cohort (n=500):

* documented negative HIV test at screening
* age >50 years at study entry
* self defined white or black African ethnicity
* registered with a General Practitioner and gives permission for contact with that General Practitioner.

Exclusion Criteria:

* in the opinion of the investigator, those unable or unwilling to comply with the requirements of the study
* life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV positive over 50 years HIV positive between 18 and 50 years HIV negative over 50 years White Black african
Sampling Method: Probability Sample
Enrollment: 1377 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Sabine, PhD, Study Director — University College, London; Alan Winston, MD, Study Director — Imperial College London
Locations (8):
- University College Dublin School of Medicine and Medical Sciences, Mater Misericordiae University Hospital, Dublin, Ireland
- United Kingdom (7):
  - Royal Sussex County Hospital, Brighton, Sussex
  - Homerton University Hospital NHS Foundation Trust, London
  - Royal Free Hospital, London
  - Kings College Hospital NHS Trust, London
  - Chelsea and Westminster Hospital, London
  - St Marys Hospital NHS Trust, London
  - University College NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Francesco D, Underwood J, Post FA, Vera JH, Williams I, Boffito M, Sachikonye M, Anderson J, Mallon PW, Winston A, Sabin CA; POPPY study group. Defining cognitive impairment in people-living-with-HIV: the POPPY study. BMC Infect Dis. 2016 Oct 28;16(1):617. doi: 10.1186/s12879-016-1970-8. PMID 27793128
- [Background] Underwood J, De Francesco D, Post FA, Vera JH, Williams I, Boffito M, Mallon PW, Anderson J, Sachikonye M, Sabin C, Winston A; Pharmacokinetic and Clinical Observations in People Over Fifty (POPPY) study group. Associations between cognitive impairment and patient-reported measures of physical/mental functioning in older people living with HIV. HIV Med. 2017 May;18(5):363-369. doi: 10.1111/hiv.12434. Epub 2016 Oct 26. PMID 27785907
- [Background] Bagkeris E, Burgess L, Mallon PW, Post FA, Boffito M, Sachikonye M, Anderson J, Asboe D, Garvey L, Vera J, Williams I, Johnson M, Babalis D, De Francesco D, Winston A, Sabin CA. Cohort profile: The Pharmacokinetic and clinical Observations in PeoPle over fiftY (POPPY) study. Int J Epidemiol. 2018 Oct 1;47(5):1391-1392e. doi: 10.1093/ije/dyy072. No abstract available. PMID 29746638
- [Background] Underwood J, De Francesco D, Leech R, Sabin CA, Winston A; Pharmacokinetic and Clinical Observations in PeoPle Over fiftY (POPPY) study. Medicalising normality? Using a simulated dataset to assess the performance of different diagnostic criteria of HIV-associated cognitive impairment. PLoS One. 2018 Apr 11;13(4):e0194760. doi: 10.1371/journal.pone.0194760. eCollection 2018. PMID 29641619
- [Background] De Francesco D, Verboeket SO, Underwood J, Bagkeris E, Wit FW, Mallon PWG, Winston A, Reiss P, Sabin CA; Pharmacokinetic and Clinical Observations in PeoPle Over fiftY (POPPY) study and the AGEhIV Cohort Study. Patterns of Co-occurring Comorbidities in People Living With HIV. Open Forum Infect Dis. 2018 Oct 24;5(11):ofy272. doi: 10.1093/ofid/ofy272. eCollection 2018 Nov. PMID 30465014
- [Background] Pool E, Winston A, Bagkeris E, Vera JH, Mallon P, Sachikonye M, Post FA, Pozniak A, Boffito M, Anderson J, Williams I, Johnson M, Burgess L, Sabin CA; Pharmacokinetic and Clinical Observations in People over Fifty (POPPY) study team. High-risk behaviours, and their associations with mental health, adherence to antiretroviral therapy and HIV parameters, in HIV-positive men who have sex with men. HIV Med. 2019 Feb;20(2):131-136. doi: 10.1111/hiv.12690. Epub 2018 Dec 12. PMID 30548745
- [Background] Halloran MO, Boyle C, Kehoe B, Bagkeris E, Mallon P, Post FA, Vera J, Williams I, Anderson J, Winston A, Sachikonye M, Sabin C, Boffito M. Polypharmacy and drug-drug interactions in older and younger people living with HIV: the POPPY study. Antivir Ther. 2019;24(3):193-201. doi: 10.3851/IMP3293. PMID 30700636
- [Background] De Francesco D, Underwood J, Bagkeris E, Boffito M, Post FA, Mallon P, Vera JH, Williams I, Anderson J, Johnson M, Sabin CA, Winston A; Pharmacokinetic and Clinical Observations in People over Fifty (POPPY) study. Depression, lifestyle factors and cognitive function in people living with HIV and comparable HIV-negative controls. HIV Med. 2019 Apr;20(4):274-285. doi: 10.1111/hiv.12714. Epub 2019 Feb 8. PMID 30734983
- [Background] De Francesco D, Winston A, Underwood J, Cresswell FV, Anderson J, Post FA, Williams I, Mallon PW, Sachikonye M, Babalis D, Vera JH, Bagkeris E, Milinkovic A, Sabin CA. Cognitive function, depressive symptoms and syphilis in HIV-positive and HIV-negative individuals. Int J STD AIDS. 2019 Apr;30(5):440-446. doi: 10.1177/0956462418817612. Epub 2019 Jan 10. PMID 30999830
- [Background] Dhillon S, Sabin CA, Alagaratnam J, Bagkeris E, Post FA, Boffito M, Anderson J, Vera J, Williams I, Johnson M, Sachikonye M, Babalis D, Mallon PW, Winston A; Pharmacokinetic and Clinical Observations in People over Fifty (POPPY) study. Level of agreement between frequently used cardiovascular risk calculators in people living with HIV. HIV Med. 2019 May;20(5):347-352. doi: 10.1111/hiv.12731. Epub 2019 Mar 14. PMID 30873751
- [Background] De Francesco D, Underwood J, Bagkeris E, Anderson J, Williams I, Vera JH, Post FA, Boffito M, Johnson M, Mallon PWG, Winston A, Sabin CA; Pharmacokinetic and Clinical Observations in PeoPle Over fiftY (POPPY) study. Risk factors and impact of patterns of co-occurring comorbidities in people living with HIV. AIDS. 2019 Oct 1;33(12):1871-1880. doi: 10.1097/QAD.0000000000002293. PMID 31259766
- [Background] Savinelli S, De Francesco D, Feeney ER, Babalis D, Bagkeris E, Post FA, Boffito M, Williams I, Vera J, Johnson M, Anderson J, Sachikonye M, Winston A, Sabin C, Mallon P. Factors associated with obesity in the Pharmacokinetic and Clinical Observations in People over Fifty (POPPY) cohort: an observational cross-sectional analysis. HIV Med. 2020 Aug;21(7):441-452. doi: 10.1111/hiv.12857. Epub 2020 Apr 20. PMID 32311831
- [Background] Wang X, Boffito M, Dickinson L, Bagkeris E, Khoo S, Post FA, Vera J, Williams I, Ndoutoumou A, Anderson J, Mallon P, McClure M, Winston A, Sabin C; POPPY Study. Plasma nucleotide reverse transcriptase inhibitor concentration and their associations with liver and renal parameters in people living with HIV. AIDS. 2020 Apr 1;34(5):790-793. doi: 10.1097/QAD.0000000000002479. PMID 32167992
- [Background] Sabin CA, Kunisaki KM, Bagkeris E, Post FA, Sachikonye M, Boffito M, Anderson J, Mallon P, Williams I, Vera JH, Johnson M, Babalis D, Winston A. Respiratory symptoms and chronic bronchitis in people with and without HIV infection. HIV Med. 2021 Jan;22(1):11-21. doi: 10.1111/hiv.12955. Epub 2020 Sep 6. PMID 32892488
- [Background] Sabin CA, Harding R, Bagkeris E, Geressu A, Nkhoma K, Post FA, Sachikonye M, Boffito M, Anderson J, Mallon PWG, Williams I, Vera J, Johnson MA, Babalis D, Winston A. The predictors of pain extent in people living with HIV. AIDS. 2020 Nov 15;34(14):2071-2079. doi: 10.1097/QAD.0000000000002660. PMID 32773481
- [Background] Winston A, De Francesco D, Post F, Boffito M, Vera J, Williams I, Anderson J, Mallon PWG, Sabin CA; POPPY Study Group. Comorbidity indices in people with HIV and considerations for coronavirus disease 2019 outcomes. AIDS. 2020 Oct 1;34(12):1795-1800. doi: 10.1097/QAD.0000000000002606. PMID 32732634
- [Result] Sabin CA, Harding R, Bagkeris E, Nkhoma K, Post FA, Sachikonye M, Boffito M, Anderson J, Mallon PWG, Williams I, Vera J, Johnson M, Babalis D, Winston A. Pain in people living with HIV and its association with healthcare resource use, well being and functional status. AIDS. 2018 Nov 28;32(18):2697-2706. doi: 10.1097/QAD.0000000000002021. PMID 30289809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV Positive Over 50 Years of Age | HIV Positive Under the Age of 50 | HIV Negative Over the Age of 50
Started | 699 | 374 | 304
Completed | 672 | 363 | 299
Not Completed | 27 | 11 | 5
Not completed — Death | 10 | 0 | 1
Not completed — Withdrawal by Subject | 17 | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Positive Over 50 Years of Age | HIV Positive Under the Age of 50 | HIV Negative Over the Age of 50 | Total
Number analyzed (Participants) | 699 | 374 | 304 | 1377
Age, Continuous [Median (Full Range); unit: years] | 57 [53 to 62] | 43 [37 to 47] | 58 [53 to 63] | 56 [53 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 72 | 109 | 268
  Male | 612 | 302 | 195 | 1109
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 96 | 75 | 31 | 202
  White | 603 | 299 | 273 | 1175
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Prevalence of Reported Aches and Pains in the Last Month Across the 3 Age Groups
Description: The number of patients reporting aches and pains in the 3 arms were used to analyse the incidence and outcomes of co-morbidities in older-HIV-positive people and their relationship with demographic/clinical factors.Comparison of three groups HIV+ve >50, HIV+<50 and HIV-ve >50.
Time Frame: after 1 year
Measure: Number; unit: participants
Groups:
- HIV Positive Over 50 Years of Age (Median Age 57); HIV Positive Under the Age of 50 (Median Age 43): All study subjects will undergo a whole body DEXA scan (dual energy X-ray absorptiometry). at the beginning and end of the study.
  Blood sample collections for the determination of the plasma concentrations of tenofovir and the third agent (i.e. a non-nucleoside reverse transcriptase, protease, entry or integrase inhibitor) in the patient's regimen will be drawn
- HIV Negative Over the Age of 50 (Median Age 58): All study subjects will undergo a whole body DEXA scan (dual energy X-ray absorptiometry). at the beginning and end of the study.
Arm/Group | HIV Positive Over 50 Years of Age (Median Age 57) | HIV Positive Under the Age of 50 (Median Age 43) | HIV Negative Over the Age of 50 (Median Age 58)
Number analyzed (Participants) | 699 | 374 | 304
participants | 473 | 224 | 188

ADVERSE EVENTS:
Time Frame: 1 year on average
Description: Given the observational and non-interventional nature of this study, the patients underwent aging assessemnt only and no additional information on SAEs was captured for the purpose of the Aging assement.
  Also, given the observational and non-interventional nature of this study, no serious, unexpected adverse drug reactions (SUSARs) reporting will be undertaken. As all subjects continue with their general clinical care, which is unaltered during the course of this study.
Groups:
- HIV Positive Under the Age of 50; HIV Positive Over 50 Years of Age: All study subjects will undergo a whole body DEXA scan (dual energy X-ray absorptiometry). at the beginning and end of the study.
  Blood sample collections for the determination of the plasma concentrations of tenofovir and the third agent (i.e. a non-nucleoside reverse transcriptase, protease, entry or integrase inhibitor) in the patient's regimen will be drawn.
  No adverse events have been reported for this group.
- HIV Negative Over the Age of 50: All study subjects will undergo a whole body DEXA scan (dual energy X-ray absorptiometry). at the beginning and end of the study.
  No adverse events have been reported for this group.
Arm/Group | HIV Positive Under the Age of 50 | HIV Negative Over the Age of 50 | HIV Positive Over 50 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/699 | 0/379 | 0/304
Serious Adverse Events (participants affected / at risk) | 0/699 | 0/379 | 0/304
Other Adverse Events (participants affected / at risk) | 0/699 | 0/379 | 0/304

LIMITATIONS AND CAVEATS:
Limitations of the POPPY study include the lack of a young HIV-negative group that would facilitate a direct comparison with the younger group of PLWH, and an over representation of white women among the HIV-negative control group. Due to time and budget constraints, this was not feasible. Future studies should consider incorporating such a group in their design in order to understand patterns and behaviours as well as similarities and differences compared with younger PLWH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT01737047/Prot_SAP_000.pdf